CLINICAL TRIAL: NCT02237586
Title: Effect of Plasmodium Falciparum Exposure and Sickle Cell Trait on Infection Rates and Kinetics After IV Administration of PfSPZ Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Centre de Recherche Médicale de Lambaréné (Other); Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LACHMI-001
Record Dates: First submitted 2014-08-27; First posted 2014-09-11 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Plasmodium Falciparum Malaria; Malaria
Keywords: Plasmodium falciparum malaria; Malaria; PfSPZ Challenge; Controlled Human Malaria Infection (CHMI); Sickle Cell Trait; Sporozoites
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Sickle Cell Trait

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group IA (Experimental): Adults with naturally acquired immunity and HbAA (Group IA, n=10)
  As any parasitemia other than PfSPZ will interfere with results, volunteers will undergo a treatment course against P. falciparum with a five-day course of 12-hourly 5 mg/kg clindamycin (corresponds to a 300 mg tablet of clindamycin base administered twice daily). This will be completed no less than three days prior to CHMI. The initial challenge dose of 3,200 PfSPZ Challenge will be administered once intravenously. If 50% or less of volunteers become parasitemic in Groups IA or IS, 10 additional volunteers will be enrolled and challenged with 12,800 PfSPZ. Effective treatment will be initiated immediately upon development of parasitemia together with the presence of symptoms associated with malaria.
  Interventions: Biological: PfSPZ Challenge
- Group IS (Experimental): Adults with naturally acquired immunity and HbAS (Group IS, n=10)
  As any parasitemia other than PfSPZ will interfere with results, volunteers will undergo a treatment course against P. falciparum with a five-day course of 12-hourly 5 mg/kg clindamycin (corresponds to a 300 mg tablet of clindamycin base administered twice daily). This will be completed no less than three days prior to CHMI. The initial challenge dose of 3,200 PfSPZ Challenge will be administered once intravenously. If 50% or less of volunteers become parasitemic in Groups IA or IS, 10 additional volunteers will be enrolled and challenged with 12,800 PfSPZ. Effective treatment will be initiated immediately upon development of parasitemia together with the presence of symptoms associated with malaria.
  Interventions: Biological: PfSPZ Challenge
- Group NI (Experimental): Adults without previous exposure to malaria and HbAA (Group NI, n=5)
  As any parasitemia other than PfSPZ will interfere with results, volunteers will undergo a treatment course against P. falciparum with a five-day course of 12-hourly 5 mg/kg clindamycin (corresponds to a 300 mg tablet of clindamycin base administered twice daily). This will be completed no less than three days prior to CHMI. The initial challenge dose of 3,200 PfSPZ Challenge administered once intravenously should lead to consistent infection in naïve adults (15/15 in prior studies) and thus should infect all volunteers in Group NI. Effective treatment will be initiated immediately upon development of parasitemia together with the presence of symptoms associated with malaria.
  Interventions: Biological: PfSPZ Challenge

INTERVENTIONS:
Biological: PfSPZ Challenge — live, aseptic, cryopreserved P. falciparum sporozoites

SUMMARY:
The study is designed to establish infectivity of Plasmodium falciparum sporozoites (PfSPZ) via intravenous (IV) administration in three groups with different malaria immunity-status:

1. Adults with a history of lifelong malaria exposure without sickle cell trait (HbAA)
2. Adults with a history of lifelong malaria exposure with sickle cell trait (HbAS)
3. Adults without previous malaria episodes without sickle cell trait (HbAA)

Initially a dose of 3,200 PfSPZ will be given and the time until thick blood smear positivity after challenge will be assessed. If in any of the groups with a history of lifelong malaria exposure, 50% or less of individuals become thick blood smear positive during the 28 days post injection of PfSPZ Challenge, the dose will be increased 4-fold to 12,800 PfSPZ in this group.

DETAILED DESCRIPTION:
LACHMI-001 is a partially-blinded, human pilot trial to study immunity against P. falciparum malaria in a controlled infection setting. The main objective is to characterise the role of sickle cell trait and naturally acquired immunity in development of malaria, defined by positive smear for P. falciparum and signs or symptoms associated with malaria. Three groups of volunteers will receive radical cure treatment and subsequently PfSPZ Challenge by IV administration. The groups are:

1. Adults with naturally acquired immunity and HbAA (Group IA, n=10-20)
2. Adults with naturally acquired immunity and HbAS (Group IS, n=10-20)
3. Adults without previous exposure to malaria and HbAA (Group NI, n=5)

The initial challenge dose of 3,200 PfSPZ administered once intravenously leads to consistent infection in naïve adults (15/15 in prior studies) and thus should infect all volunteers in Group 3. However, volunteers with naturally acquired immunity or sickle cell trait might require a higher dose. Thus if 50% or less of volunteers become parasitemic in Groups IA or IS, 10 additional volunteers will be enrolled and challenged with 12,800 PfSPZ. All volunteers will be healthy adults aged 18 to 30 years. Safety and infectivity data will be collected for each of the regimens and dose-levels. Effective treatment is initiated immediately upon development of parasitemia together with the presence of symptoms associated with malaria.

Laboratory staff reading blood films and processing samples will be blinded to group allocation. Volunteers and clinical investigators will be blinded to group allocation among the IA and IS groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 30 years
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Women only: must agree to practice continuous effective contraception for the duration of the study (a method which results in a low failure rate; i.e. less than 1% per year)
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local blood banking eligibility criteria
* Written informed consent to undergo CHMI
* Reachable (24/7) by mobile phone during the whole study period
* Willingness to take two curative anti-malarial regimens
* Agreement to stay overnight for observation during the period of intensive follow-up post-challenge if required
* Answer all questions on the informed consent quiz correctly
* A body mass index < 35
* A haemoglobin concentration ≥10 g/dl for women and ≥12 g/dl for men

Additional inclusion criteria for IA and IS group only:

- History of long term residence (>10 years) in area known to have significant transmission of P. falciparum -

Exclusion Criteria:

* Use of anti-malarials within 30 days of study enrolment
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrolment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin)
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period
* Prior receipt of an investigational malaria vaccine
* Immunization with more than 1 other vaccines within the past month.
* HIV infection
* Hemoglobin SS
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment
* Pregnancy, lactation or intention to become pregnant during the study
* A history of allergic disease or reactions likely to be exacerbated by malaria
* Contraindications to the use of the first-line anti-malarial medications: artemether/lumefantrine or atovaquone/proguanil.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the study
* History of epileptic seizures
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60 g (men) or 40 g (women) per day
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Falling in moderate risk or higher categories for fatal or non-fatal cardiovascular event within 5 years (>10%) determined by non-invasive criteria for cardiac risk
* Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial contractions, right of left bundle branch block, advanced A-V heart block (secondary or tertiary)
* A QT/QTc interval > 450 ms
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination
* Any other significant disease, disorder or finding which, in the opinion of the Investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Additional exclusion criteria for NI group only:

* History of P. falciparum malaria
* History of long term residence (>5 years) in area known to have significant transmission of P. falciparum
* Presence of sickle cell trait
* Known thalassemia or thalassemia trait

Exclusion Criterion on Day of Challenge or Day before Challenge

* Acute disease, defined as moderate or severe illness with or without fever
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Days from inoculation to start of malaria episode | From day of injection until day 28
  The time from parasite inoculation to first detection of malaria will be assessed by thick blood film microscopy and a clinical questionnaire. Malaria is defined as both parasitemia and clinical symptoms suggestive of malaria.
Frequency, incidence and nature of adverse events | From day of injection until day 28
  The safety of PfSPZ Challenge administered IV and the resultant P. falciparum infection will be assessed by analysing actively and passively collected data from clinical review of volunteers and laboratory measurements.

SECONDARY OUTCOMES:
Dynamics of P. falciparum parasite growth | From day 6 after injection until approximately day 28
  The dynamics of P. falciparum parasite growth following administration of PfSPZ Challenge is assessed by analyzing parasite multiplication rates using highly sensitive qPCR for P. falciparum DNA. Measurements will be used to model parasite kinetics and to estimate the number of infected liver cells.

OTHER OUTCOMES:
Cellular and humoral immune responses against parasites | From screening until 6 months
  Cellular and humoral immune responses against parasites will be assessed by individual and collective results of cytometry, enzyme-linked immunospot analysis (ELISpot), enzyme-linked immunosorbent assay (ELISA), immunofluorescence assay (IFA), inhibition of sporozoite invasion of hepatocytes assay (ISI), quantification of erythrophagocytosis, B-cell typing and isolation as well as protein microarray.
Stage specific expression patterns of parasite genes | From screening until 6 months
  Stage specific expression patterns of parasite genes will be assessed by RNA quantification using reverse transcriptase PCR (rtPCR) and transcriptional profiling on microarray and sequencing platforms. Differences in miRNA expression between AA and AS erythrocytes will be determined and related to multiplication rates.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lell, MD, Principal Investigator — Centre de Recherche Médicale de Lambaréné
Locations (1):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Gabon

REFERENCES:
- [Derived] Requena P, Gomez-Perez GP, McCall MBB, Barrios D, Aguilar R, Fernandez-Morata J, Vidal M, Campo JJ, Sanchez C, Yazdabankhsh M, Sim BKL, Hoffman SL, Kremsner P, Lell B, Mordmuller B, Dobano C, Moncunill G. Effect of controlled human Plasmodium falciparum infection on B cell subsets in individuals with different levels of malaria immunity. Med Microbiol Immunol. 2025 Sep 27;214(1):47. doi: 10.1007/s00430-025-00847-x. PMID 41014333